CLINICAL TRIAL: NCT05049967
Title: iKnow: A Prospective Study to Evaluate the Use of Multi-omics in Multi-System, Early Onset Disorders
Acronym: iKnow
Status: Active, not recruiting | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: ILMN-iKnow
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Outpatient setting with eighty percent consisting of prior negative genome cases that have previously received a clinical whole genome sequencing (cWGS) test. Remaining twenty percent will be positive controls who previously have a definitive diagnosis from clinical genetic testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study to further understand the value that a multi-omic approach has in individuals with a multi system, early onset disorder that does not have a molecular diagnosis by whole genome sequencing.

DETAILED DESCRIPTION:
Understand the value and utilization of integrated multi-omics, in multi-system early onset disorders that have failed to yield findings by whole genome sequencing

ELIGIBILITY:
Inclusion Criteria:

* Undiagnosed probands must meet all of the following:

  1. Must be able to understand and sign an informed consent and speak, read, and write in their native language (if the subject is a minor, their parent must have these abilities)
  2. Proband between the ages of 12 months and 65 years
  3. Study consent and participation of at least two unaffected family members (biological parents preferred. One biological parent and unaffected sibling allowed)
  4. If applicable, unaffected sibling must be between the ages of 12 months and 65 years
  5. A high prior probability of a multi-system early onset undiagnosed genetic disorder based on an expert medical assessment
  6. Clinical WGS that did not yield a definitive diagnosis
  7. It is preferred but not required that ancestry is from an under-represented population in current clinical genetic and translational research data repositories, especially African American, Asian American and Native American
  8. Must be willing to have blood, urine and fecal samples taken to include participating family members

Diagnosed probands must meet all of the following:

1. Must be able to understand and sign an informed consent and speak, read, and write in their native language (if the subject is a minor, its Parent or Legally Authorized Representative must have these abilities).
2. Proband between the ages of 12 months and 65 years
3. Study consent and participation of at least two unaffected family members (biological parents preferred. One biological parent and unaffected sibling allowed)
4. If applicable, unaffected sibling must be between the ages of 12 months and 65 years
5. Known genetic cause(s) of disease, disorder, or phenotypic defect through prior clinical whole genome sequencing
6. It is preferred but not required that ancestry is from an under-represented population in current clinical genetic and translational research data repositories, especially African American, Asian American and Native American
7. Must be willing to have blood, urine and fecal samples taken to include participating family members

Exclusion Criteria:

* Undiagnosed probands must not meet any:

  1. Known non-genetic cause(s) of disease, disorder, or phenotypic defect
  2. Principal Investigator decides that the study is not in the best interest of the proband

Diagnosed probands must not meet any:

1. Principal Investigator decides that the study is not in the best interest of the proband

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient setting with eighty percent consisting of prior negative genome cases that have previously received a clinical whole genome sequencing (cWGS) test. Remaining twenty percent will be positive controls who previously have a definitive diagnosis from clinical genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Based on analysis of data from completed clinical utility evaluation surveys following receipt of study results by the PI, assess whether a patient's change of management resulted from the multi-omic results | 120 Days
  Understand the value and utilization of integrated multi-omics, in multi-system early onset disorders that have failed to yield findings by whole genome sequencing

SECONDARY OUTCOMES:
Number of diagnoses yielded by each of the different orthogonally confirmed assay results | 120 Days
  Assess the number of new diagnoses yielded by each approach
Analyze data from completed clinical utility evaluation surveys; number of patients with change of management and whether the change was due to a diagnosis yielded by multiomic results | 120 Days
  Analyze the clinical utility derived from a diagnosis
Data utilization of multi-omic dataset for scientific community | 120 Days
  Establish a multi-omic reference dataset from resource limited populations that can be used by the scientific community

CONTACTS AND LOCATIONS:
Overall Officials: Ali Crawford, PhD, Study Director — Illumina, Inc.
Locations (1):
- Clinic for Special Children, Strasburg, Pennsylvania, United States